CLINICAL TRIAL: NCT00146614
Title: Tacrolimus, Sirolimus and Methotrexate as Graft Versus Host Disease Prophylaxis After Allogeneic Non-Myeloablative Peripheral Blood Stem Cell Transplantation
Brief Title: Tacrolimus, Sirolimus and Methotrexate as Graft Versus Host Disease Prophylaxis After Blood Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Edwin P. Alyea, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-057
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Graft Versus Host Disease; Hematologic Malignancies
Keywords: Graft versus Host Disease; GVHD; Stem Cell Transplantation; Tacrolimus; Sirolimus; Methotrexate; allogeneic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — Sirolimus; Tacrolimus; Methotrexate; Stem Cell Transplantation

INTERVENTIONS:
Drug: Sirolimus
Drug: Tacrolimus
Drug: Methotrexate
Procedure: Stem Cell Transplantation

SUMMARY:
The purpose of this study is to determine if the incidence of Graft vs. Host Disease (GVHD) after non-myeloablative transplantation can be reduced by using a combination of three immune suppressive medication; sirolimus, tacrolimus and methotrexate.

DETAILED DESCRIPTION:
* Patients will be admitted to the hospital and receive chemotherapy and stem cell transplant(SCT). The total duration of hospitalization for the procedure is approximately 8 days. Once admitted the patient will receive fludarabine daily for 4 days, busulfex once daily for 4 days. Two days after chemotherapy has ended, the patient will receive the infusion of donor cells.
* Just prior to the transplant and following the transplant, patients will receive sirolimus (orally), tacrolimus (orally) and low doses of methotrexate (chemotherapy). Methotrexate will be given on days 1,3 and 6 after transplant.
* Sirolimus will be tapered beginning week 9 after transplant if there is no evidence of GVHD and will be eliminated on week 26 if clinically feasible.
* Tacrolimus will be tapered beginning week 9 after transplant if there is no evidence of GVHD and will be eliminated on week 26 if clinically feasible.
* Patients will also receive medication to help prevent possible infection.
* After stem cell infusion, patients will be examined and have blood tests weekly for 1 month. At the 1 month visit, a bone marrow biopsy will performed looking for evidence of donor cells in the bone marrow. After the one month evaluation the patient will be examined every 2 weeks and a repeat bone marrow performed 3-4 months after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies who are at a high risk of complications after conventional transplantation.
* Donors (both related and unrelated) who are identical at 6 HLA loci.
* Age greater than 18
* ECOG Performance Status 0-2
* Life expectancy of greater than 100 days.

Exclusion Criteria:

* Pregnancy
* Evidence of HIV infection
* Heart failure uncontrolled by medications
* Total Bilirubin > 2.0mg/dl due to hepatocellular dysfunction
* AST > 90
* Serum creatinine > 2.0
* Cholesterol > 300 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105
Dates: Start 2002-07; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
To assess the effect on the incidence and severity of GVHD by adding sirolimus, tacrolimus and methotrexate to GVHD prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin P. Alyea, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts